CLINICAL TRIAL: NCT04138056
Title: A Phase II Study of a Primary Dose of Investigational RSV Maternal Vaccine, Given Alone or With Boostrix, With a 2nd Dose Investigational RSV Maternal Vaccine
Brief Title: A Study of a Vaccine Against Respiratory Syncytial Virus (RSV) When Given Alone and Together With a Vaccine Against Diphtheria, Pertussis and Tetanus (Tdap) Viruses Followed by a 2nd Dose of the RSV Vaccine to Healthy Non-Pregnant Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 209141; 2019-002258-22 (EudraCT Number)
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Results first posted 2022-12-19 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data will be collected in an observer-blind manner. In an observer-blind study, the subject and the site and sponsor personnel involved in the clinical evaluation of the subjects are blinded while other study personnel may be aware of the treatment assignment. By observer-blind, it is meant that during the course of the study, the vaccine(s) recipient and those responsible for the evaluation of any study endpoint (e.g. safety, reactogenicity) will all be unaware of which vaccines were administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- RSV120_dTpa_RSV120(Pooled) (Experimental): Subjects received one dose of 120 μg RSVPreF3 formulation 3 vaccine and either one dose of 300 μg or 500 μg dTpa (Boostrix) vaccine on Day 1 of the Primary Study and were followed up until Day 181. The subjects that agreed to participate in the Extension Study received a second dose of 120 μg RSVPreF3 formulation 3 vaccine 12 to 18 months post 1st vaccination and were followed up until the study end.
  Interventions: Biological: RSVPreF3 formulation 3; Biological: Boostrix-ex-US; Biological: Boostrix-US
- RSV120_Placebo_RSV120(Pooled) (Placebo Comparator): Subjects received one dose of 120 μg RSVPreF3 formulation 3 vaccine and one dose of Placebo on Day 1 of the Primary Study and were followed up until Day 181. The subjects that agreed to participate in the Extension Study received a second dose of 120 μg RSVPreF3 formulation 3 vaccine 12 to 18 months post 1st vaccination and were followed up until the study end.
  Interventions: Biological: RSVPreF3 formulation 3; Drug: Placebo
- RSV60_dTpa_RSV120(Pooled) (Experimental): Subjects received one dose of 60 μg RSVPreF3 formulation 2 vaccine and either one dose of 300 μg or 500 μg dTpa vaccine on Day 1 of the Primary Study and were followed up until Day 181. The subjects that agreed to participate in the Extension Study received one dose of 120 μg RSVPreF3 formulation 3 vaccine 12 to 18 months post 1st vaccination and were followed up until the study end.
  Interventions: Biological: RSVPreF3 formulation 3; Biological: RSVPreF3 formulation 2; Biological: Boostrix-ex-US; Biological: Boostrix-US
- RSV60_Placebo_RSV120(Pooled) (Placebo Comparator): Subjects received one dose of 60 μg RSVPreF3 formulation 2 vaccine and one dose of Placebo on Day 1 of the Primary Study and were followed up until Day 181. The subjects that agreed to participate in the Extension Study received one dose of 120 μg RSVPreF3 formulation 3 vaccine 12 to 18 months post 1st vaccination and were followed up until the study end.
  Interventions: Biological: RSVPreF3 formulation 3; Biological: RSVPreF3 formulation 2; Drug: Placebo
- dTpa_Placebo_RSV120(Pooled) (Placebo Comparator): Subjects received one dose of Placebo and either one dose of 300 μg or 500 μg dTpa vaccine on Day 1 of the Primary Study and were followed up until Day 181. The subjects that agreed to participate in the Extension Study received one dose of 120 μg RSVPreF3 formulation 3 vaccine 12 to 18 months post 1st vaccination and were followed up until the study end.
  Interventions: Biological: RSVPreF3 formulation 3; Biological: Boostrix-ex-US; Biological: Boostrix-US; Drug: Placebo

INTERVENTIONS:
Biological: RSVPreF3 formulation 3 — One dose of RSVPreF3 formulation 3 vaccine administered intramuscularly in the left or in the non-dominant arm.
Biological: RSVPreF3 formulation 2 — One dose of RSVPreF3 formulation 2 vaccine administered intramuscularly in the left arm.
  Arms: RSV60_Placebo_RSV120(Pooled); RSV60_dTpa_RSV120(Pooled)
Biological: Boostrix-ex-US — One dose of the dTpa (Ex-US formulation) vaccine administered intramuscularly in the right arm.
  Arms: RSV120_dTpa_RSV120(Pooled); RSV60_dTpa_RSV120(Pooled); dTpa_Placebo_RSV120(Pooled)
Biological: Boostrix-US — One dose of the dTpa vaccine (US formulation) administered intramuscularly in the right arm.
  Arms: RSV120_dTpa_RSV120(Pooled); RSV60_dTpa_RSV120(Pooled); dTpa_Placebo_RSV120(Pooled)
Drug: Placebo — One dose of placebo (NaCl solution) administered intramuscularly in either the left or the right arm.
  Arms: RSV120_Placebo_RSV120(Pooled); RSV60_Placebo_RSV120(Pooled); dTpa_Placebo_RSV120(Pooled)

SUMMARY:
The purpose of this study is to evaluate the safety, ability of GSK Biologicals' investigational RSV maternal vaccine (RSVPreF3) to generate an immune response and the degree to which the vaccine can cause side effects, when administered alone and in combination with Boostrix vaccine in healthy non-pregnant women 18-45 years of age. Two dose levels of RSVPreF3 and 2 Boostrix [Diphtheria, Tetanus and acellular Pertussis (dTpa) vaccine] formulations (US and ex-US) will be evaluated. A 2nd dose of RSVPreF3 will be administered in an extension of the study to assess the durability of the immune response after the first dose vaccination, and to assess the safety and immunogenicity following a second dose vaccination of the RSVPreF3 maternal vaccine.

ELIGIBILITY:
Inclusion Criteria:

Primary study

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the subject prior to performance of any study specific procedure.
* Healthy female subjects; as established by medical history and clinical examination, aged 18 to 45 years at the time of the 1st vaccination;
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to primary vaccination, and
  * has a negative pregnancy test on the day of primary vaccination, and
  * has agreed to continue adequate contraception for 90 days after completion of the vaccination.
* No local condition precluding injection in both left and right deltoid muscles.

Extension study

* Completed primary study and received 1st dose of a study vaccine.
* Written or witnessed/thumb printed informed consent obtained from the subject prior to performance of any study specific procedure to the study extension.

All subjects must satisfy ALL the following criteria:

* Subjects who can and will comply with the requirements of the protocol.
* Female subjects remain healthy; as established by medical history and clinical examination, aged 18 to 45 years at the time of the 1st vaccination;
* Female subjects of childbearing potential are eligible for the extension, if the subject:

  * has practiced adequate contraception for 30 days prior to 2nd vaccination
  * has a negative pregnancy test with results available on the day of 2nd vaccination
  * has agreed to continue adequate contraception for 90 days after completion of the 2nd vaccination.

Exclusion Criteria:

Primary study

Medical conditions

* History of any reaction/hypersensitivity likely to be exacerbated by any vaccines' component;
* Any confirmed/suspected immunosuppressive/immunodeficient condition, based on medical history and physical examination;
* Hypersensitivity to latex;
* Major congenital defects;
* Acute/chronic clinically significant pulmonary, cardiovascular, hepatic/renal functional abnormality;
* Significant/uncontrolled psychiatric illness;
* Recurrent history/uncontrolled neurological disorders/seizures;
* Documented HIV-positive subject;
* History of/current autoimmune disease;
* Body mass index (BMI)>40 kg/m^2;
* Any clinically significant hematological parameter and/or biochemical laboratory abnormality.
* Any other clinical condition that might pose additional risk to the subject due to participation in the study.

Prior/Concomitant therapy

* Use of any investigational/non-registered product other than the study vaccines during the period starting 30 days before 1st vaccination, or planned use during the study;
* Administration of long-acting immune-modifying drugs at any time during the study;
* Administration of immunoglobulins and/or any blood products/plasma derivatives during the period starting 3 months before the 1st vaccination or planned administration during the study;
* Chronic administration of immunosuppressants/other immune-modifying drugs during the period starting 3 months prior to 1st vaccine dose(s). For corticosteroids, this will mean prednisone ≥5 mg/day, or equivalent. Inhaled and topical steroids are allowed;
* Planned administration/administration of a vaccine not foreseen by the study protocol within the period starting 30 days before and ending 30 days after study 1st vaccination, with the exception of any licensed influenza vaccine which may be administered ≥ 15 days before/after study vaccination;
* Administration of a vaccine containing diphtheria, tetanus/pertussis antigens/diphtheria and tetanus toxoids within the previous 5 years;
* Previous experimental vaccination against RSV;

Prior/Concurrent clinical study experience • Concurrently participating in another clinical study, at any time during the study, in which the subject has been/will be exposed to an investigational/a non-investigational vaccine/product;

Other exclusions

* Pregnant/lactating female;
* Female planning to become pregnant/planning to discontinue contraceptive precautions;
* History of alcoholism, drug abuse and/or use disorder within the past 2 years;
* Any study personnel/their immediate dependents, family/household members.

Extension study

Medical conditions

* History of any reaction/hypersensitivity likely to be exacerbated by any component of the vaccines;
* Any confirmed/suspected immunosuppressive/immunodeficient condition, based on medical history and physical examination;
* Hypersensitivity to latex;
* Acute/chronic clinically significant pulmonary, cardiovascular, hepatic/renal functional abnormality;
* Significant/uncontrolled psychiatric illness;
* Recurrent history/uncontrolled neurological disorders/seizures;
* Documented HIV-positive subject;
* History of/current autoimmune disease;
* BMI>40 kg/m^2;
* Participants who experienced any SAE judged to be possibly or probably related to 1st dose of RSVPreF3, including hypersensitivity reactions.
* Any other clinical condition that might pose additional risk to the subject due to participation in the study.

Prior/Concomitant therapy

* Use of any investigational/non-registered product other than the study vaccines during the period starting 30 days before the 2nd vaccination, or planned use during the 6-month study extension;
* Administration of long-acting immune-modifying drugs at any time during the study;
* Administration of immunoglobulins and/or any blood products/plasma derivatives during the period starting 3 months before the 1st dose of study vaccines/planned administration during the study;
* Chronic administration of immunosuppressants or other immune-modifying drugs during the starting 3 months prior to the 1st vaccine dose(s). For corticosteroids, this will mean prednisone ≥5 mg/day, or equivalent. Inhaled and topical steroids are allowed;
* Planned administration/administration of a vaccine not foreseen by the study protocol within the period starting 30 days before and ending 30 days after study 2nd vaccination, with the exception of any licensed influenza vaccine which may be administered ≥ 15 days before/after study vaccination.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study, in which the subject has been/will be exposed to an investigational/a non-investigational vaccine/product;

Other exclusions

* Pregnant/lactating female at the time of Visit 4;
* Female planning to become pregnant/planning to discontinue contraceptive precautions;
* History of alcoholism, drug abuse and/or use disorder within the past 2 years;
* Any study personnel/their immediate dependents, family/household members.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 509 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (4):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Seattle, Washington
- Belgium (2):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
- Canada (2):
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, London, Ontario

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data (IPD) and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Hermida N, Ferguson M, Leroux-Roels I, Pagnussat S, Yaplee D, Hua N, van den Steen P, Anspach B, Dieussaert I, Kim JH. Safety and Immunogenicity of Respiratory Syncytial Virus Prefusion Maternal Vaccine Coadministered With Diphtheria-Tetanus-Pertussis Vaccine: A Phase 2 Study. J Infect Dis. 2024 Aug 16;230(2):e353-e362. doi: 10.1093/infdis/jiad560. PMID 38133639

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data reported in the participant flow, baseline characteristics and the immunogenicity outcome measures of the Extension Study were only analyzed for pooled groups [RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled) & dTpa_Placebo_RSV120(Pooled)], as the two formulations of dTpa vaccine (containing 300 micrograms(μg) or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies.
Period: Primary Study
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Started | 101 | 101 | 103 | 102 | 102
Completed | 95 | 93 | 100 | 100 | 98
Not Completed | 6 | 8 | 3 | 2 | 4
Not completed — Lost to Follow-up | 3 | 4 | 1 | 1 | 4
Not completed — ELIGIBILITY CRITERIA NOT FULFILLED (INCLUSION AND EXCLUSION CRITERIA) | 3 | 4 | 2 | 1 | 0
Period: Extension Study
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Started | 39 (Out of 95 subjects who completed the Primary Study, 56 subjects did not participate in the Extension Study due to non-compliance of protocol requirements (e.g. completion of the diary card, return for follow-up visits, no willingness/no informed consent obtained).) | 41 (Out of 93 subjects, who completed the Primary Study, 52 subjects did not participate in the Extension Study due to non-compliance of protocol requirements (e.g. completion of the diary card, return for follow-up visits, no willingness/no informed consent obtained).) | 46 (Out of 100 subjects, who completed the Primary Study, 54 subjects did not participate in the Extension Study due to non-compliance of protocol requirements (e.g. completion of the diary card, return for follow-up visits, no willingness/no informed consent obtained).) | 41 (Out of 100 subjects, who completed the Primary Study, 59 subjects did not participate in the Extension Study due to non-compliance of protocol requirements (e.g. completion of the diary card, return for follow-up visits, no willingness/no informed consent obtained).) | 46 (Out of 98 subjects, who completed the Primary Study, 52 subjects did not participate in the Extension Study due to non-compliance of protocol requirements (e.g. completion of the diary card, return for follow-up visits, no willingness/no informed consent obtained).)
Completed | 38 | 39 | 45 | 41 | 45
Not Completed | 1 | 2 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 2 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled) | Total
Number analyzed (Participants) | 101 | 101 | 103 | 102 | 102 | 509
Age, Customized [Mean (Standard Deviation); unit: Years] — Age, Primary Study
  Years | 31.4 (7.6) | 31.0 (8.0) | 30.8 (8.4) | 30.5 (8.3) | 30.4 (7.9) | 30.8 (8.0)
Age, Customized [Mean (Standard Deviation); unit: Years] — Population: Age, Extension Study
  Years
    number analyzed (Participants) | 39 | 41 | 46 | 41 | 46 | 213
    (all) | 32.1 (7.9) | 31.7 (8.4) | 30.4 (8.6) | 30.3 (8.4) | 32.6 (8.2) | 31.4 (8.3)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex/Gender, Primary Study
  Participants
    Female | 101 | 101 | 103 | 102 | 102 | 509
    Male | 0 | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Sex/Gender, Extension Study
  Participants
    Female: number analyzed (Participants) | 39 | 41 | 46 | 41 | 46 | 213
    Female | 39 | 41 | 46 | 41 | 46 | 213
    Male: number analyzed (Participants) | 39 | 41 | 46 | 41 | 46 | 213
    Male | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/Ethnicity, Primary Study
  Participants
    AMERICAN INDIAN OR ALASKA NATIVE | 3 | 0 | 1 | 1 | 0 | 5
    ASIAN | 1 | 3 | 2 | 4 | 4 | 14
    BLACK OR AFRICAN AMERICAN | 4 | 6 | 8 | 3 | 4 | 25
    OTHER Not specified | 2 | 2 | 2 | 2 | 3 | 11
    WHITE | 91 | 90 | 90 | 92 | 91 | 454
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race/Ethnicity, Extension Study
  Participants
    AMERICAN INDIAN OR ALASKA NATIVE: number analyzed (Participants) | 39 | 41 | 46 | 41 | 46 | 213
    AMERICAN INDIAN OR ALASKA NATIVE | 1 | 0 | 0 | 0 | 0 | 1
    ASIAN: number analyzed (Participants) | 39 | 41 | 46 | 41 | 46 | 213
    ASIAN | 1 | 0 | 1 | 2 | 0 | 4
    BLACK OR AFRICAN AMERICAN: number analyzed (Participants) | 39 | 41 | 46 | 41 | 46 | 213
    BLACK OR AFRICAN AMERICAN | 0 | 0 | 1 | 0 | 1 | 2
    OTHER Not specified: number analyzed (Participants) | 39 | 41 | 46 | 41 | 46 | 213
    OTHER Not specified | 1 | 0 | 2 | 0 | 1 | 4
    WHITE: number analyzed (Participants) | 39 | 41 | 46 | 41 | 46 | 213
    WHITE | 36 | 41 | 42 | 39 | 44 | 202

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Any Solicited Local Adverse Event (AEs) [Primary Study]
Description: Assessed solicited local AEs are: erythema, pain and swelling. Any = occurrence of the adverse event regardless of intensity grade. Any erythema and swelling = adverse event reported with a surface diameter greater than 0 millimeters.
  The analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies. The objective of this endpoint was to analyze the impact of the co-administration of RSVPreF3 with dTpa (Boostrix) (both formulations together) on the safety response to RSVPreF3.
Time Frame: From Day 1 to Day 8
Population: The analysis was performed on the Solicited Safety Set (SSS) - Primary Study which consisted of all subjects from the Exposed set (ES) - Primary Study for whom solicited safety data were available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 101 | 100 | 103 | 102 | 99
Percentage of participants
  RSVPreF3 (Left Arm), Erythema | 5.9 [2.2 to 12.5] | 5 [1.6 to 11.3] | 5.8 [2.2 to 12.2] | 5.9 [2.2 to 12.4] | 0 [0 to 3.7]
  RSVPreF3 (Left Arm), Pain | 51.5 [41.3 to 61.6] | 54 [43.7 to 64] | 52.4 [42.4 to 62.4] | 58.8 [48.6 to 68.5] | 19.2 [12 to 28.3]
  RSVPreF3 (Left Arm), Swelling | 2 [0.2 to 7] | 7 [2.9 to 13.9] | 2.9 [0.6 to 8.3] | 4.9 [1.6 to 11.1] | 0 [0 to 3.7]
  dTpa (Right Arm), Erythema | 4 [1.1 to 9.8] | 1 [0 to 5.4] | 4.9 [1.6 to 11] | 1 [0 to 5.3] | 6.1 [2.3 to 12.7]
  dTpa (Right Arm), Pain | 81.2 [72.2 to 88.3] | 25 [16.9 to 34.7] | 76.7 [67.3 to 84.5] | 18.6 [11.6 to 27.6] | 78.8 [69.4 to 86.4]
  dTpa (Right Arm), Swelling | 5 [1.6 to 11.2] | 0 [0 to 3.6] | 1.9 [0.2 to 6.8] | 1 [0 to 5.3] | 4 [1.1 to 10]

2. Primary Outcome: Percentage of Subjects With Any Solicited General AEs [Primary Study]
Description: Assessed solicited general AEs are: fatigue, gastrointestinal symptoms, headache and fever (body temperature ≥ 38 degree celcius/100.4 degree Farenhit). Any = occurrence of the adverse event regardless of intensity grade or relation to study vaccination.
  The analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies. The objective of this endpoint was to analyze the impact of the co-administration of RSVPreF3 with dTpa (Boostrix) (both formulations together) on the safety response to RSVPreF3.
Time Frame: From Day 1 to Day 8
Population: The analysis was performed on the SSS - Primary Study which consisted of all subjects from the ES - Primary Study for whom solicited safety data were available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 101 | 101 | 103 | 102 | 99
Percentage of participants
  Fatigue | 40.6 [30.9 to 50.8] | 39.6 [30 to 49.8] | 37.9 [28.5 to 48] | 32.4 [23.4 to 42.3] | 38.4 [28.8 to 48.7]
  Gastrointestinal symptoms | 23.8 [15.9 to 33.3] | 28.7 [20.1 to 38.6] | 27.2 [18.9 to 36.8] | 28.4 [19.9 to 38.2] | 28.3 [19.7 to 38.2]
  Headache | 44.6 [34.7 to 54.8] | 45.5 [35.6 to 55.8] | 35 [25.8 to 45] | 39.2 [29.7 to 49.4] | 37.4 [27.9 to 47.7]
  Temperature | 2 [0.2 to 7] | 4 [1.1 to 9.8] | 2.9 [0.6 to 8.3] | 3.9 [1.1 to 9.7] | 7.1 [2.9 to 14]

3. Primary Outcome: Percentage of Subjects With Any Unsolicited AEs [Primary Study]
Description: An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is to be reported as an unsolicited AE.
  The analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies. The objective of this endpoint was to analyze the impact of the co-administration of RSVPreF3 with dTpa (Boostrix) (both formulations together) on the safety response to RSVPreF3.
Time Frame: From Day 1 to Day 31
Population: The analysis was performed on the ES - Primary Study which consisted of all subjects who received at least 1 dose of the study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 101 | 101 | 103 | 102 | 102
Percentage of participants | 38.6 [29.1 to 48.8] | 34.7 [25.5 to 44.8] | 33 [24.1 to 43] | 37.3 [27.9 to 47.4] | 32.4 [23.4 to 42.3]

4. Primary Outcome: Number of Subjects With Any SAEs [Primary Study]
Description: A SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization or results in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study subject. Any is defined as any occurrence of SAE regardless of intensity grade or relation to study vaccination.
  The analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies. The objective of this endpoint was to analyze the impact of the co-administration of RSVPreF3 with dTpa (Boostrix) (both formulations together) on the safety response to RSVPreF3.
Time Frame: From Day 1 to Day 31
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 101 | 101 | 103 | 102 | 102
Participants | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Percentage of Subjects With Any Solicited Local AEs [Extension Study]
Description: Assessed solicited local AEs are: erythema, pain and swelling. Any = occurrence of the adverse event regardless of intensity grade. Any erythema and swelling = adverse event reported with a surface diameter greater than 0 millimeters.
  The analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies.The objective of this endpoint was to analyze the impact of the co-administration of RSVPreF3 with dTpa (Boostrix) (both formulations together) on the safety response to RSVPreF3.
Time Frame: From the Day of 2nd vaccination to Day 8 post 2nd vaccination
Population: The analysis was performed on the SSS - Extension Study which consisted of all subjects from the ES - Extension Study for whom solicited safety data were available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 39 | 39 | 46 | 41 | 44
Percentage of participants
  Erythema | 17.9 [7.5 to 33.5] | 10.3 [2.9 to 24.2] | 8.7 [2.4 to 20.8] | 14.6 [5.6 to 29.2] | 2.3 [0.1 to 12]
  Pain | 87.2 [72.6 to 95.7] | 87.2 [72.6 to 95.7] | 80.4 [66.1 to 90.6] | 85.4 [70.8 to 94.4] | 38.6 [24.4 to 54.5]
  Swelling | 12.8 [4.3 to 27.4] | 7.7 [1.6 to 20.9] | 8.7 [2.4 to 20.8] | 4.9 [0.6 to 16.5] | 2.3 [0.1 to 12]

6. Primary Outcome: Percentage of Subjects Any Solicited General AEs [Extension Period]
Description: Assessed solicited general AEs are: fatigue, gastrointestinal symptoms, headache and fever(body temperature ≥ 38 degree celcius/100.4 degree Farenhit). Any = occurrence of the adverse event regardless of intensity grade or relation to study vaccination.
  The analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies. The objective of this endpoint was to analyze the impact of the co-administration of RSVPreF3 with dTpa (Boostrix) (both formulations together) on the safety response to RSVPreF3.
Time Frame: From the Day of 2nd vaccination to Day 8 post 2nd vaccination
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 39 | 39 | 46 | 41 | 44
Percentage of participants
  Fatigue | 25.6 [13 to 42.1] | 33.3 [19.1 to 50.2] | 37 [23.2 to 52.5] | 46.3 [30.7 to 62.6] | 34.1 [20.5 to 49.9]
  Gastrointestinal symptoms | 10.3 [2.9 to 24.2] | 20.5 [9.3 to 36.5] | 15.2 [6.3 to 28.9] | 24.4 [12.4 to 40.3] | 13.6 [5.2 to 27.4]
  Headache | 28.2 [15 to 44.9] | 33.3 [19.1 to 50.2] | 32.6 [19.5 to 48] | 56.1 [39.7 to 71.5] | 31.8 [18.6 to 47.6]
  Temperature | 0 [0 to 9] | 0 [0 to 9] | 2.2 [0.1 to 11.5] | 9.8 [2.7 to 23.1] | 2.3 [0.1 to 12]

7. Primary Outcome: Percentage of Subjects With Any Unsolicited AEs [Extension Period]
Description: as for outcome 3
Time Frame: From the Day of 2nd vaccination to Day 31 post 2nd vaccination
Population: The analysis was performed on ES - Extension Study which consisted of all subjects who received at least 2 doses of the study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 39 | 41 | 46 | 41 | 46
Percentage of participants | 18 [8 to 34] | 20 [9 to 35] | 20 [9 to 34] | 29 [16 to 46] | 20 [9 to 34]

8. Primary Outcome: Number of Subjects With Any SAEs [Extension Period]
Description: as for outcome 4
Time Frame: From the Day of 2nd vaccination to Day 31 post 2nd vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 39 | 41 | 46 | 41 | 46
Participants | 0 | 0 | 0 | 1 | 0

9. Primary Outcome: RSV A Neutralizing Antibody Geometric Mean Titers (GMTs) at Screening [Primary Study]
Description: Serological assays for the determination of antibodies against RSV-A were performed by neutralization assay and titers are expressed in ED60 (Estimated Dilution 60).
  The analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies. The objective of this endpoint was to analyze the impact of the co-administration of RSVPreF3 with dTpa (Boostrix) (both formulations together) on the immunogenicity response to RSVPreF3.
Time Frame: At Screening (Day -7 to Day 1)
Population: The analysis was performed on the Per Protocol Set (PPS) - Primary Study which consisted of all subjects from the ES - Primary Study, who complied with protocol defined procedures and for whom immunogenicity results were available for the specified assay and time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 100 | 100 | 103 | 102 | 102
Titers (ED60) | 875 [745 to 1027] | 1022 [856 to 1222] | 1135 [959 to 1342] | 771 [673 to 883] | 1050 [896 to 1231]

10. Primary Outcome: RSV A Neutralizing Antibody GMTs at Day 8 [Primary Study]
Description: Serological assays for the determination of antibodies against RSV-A were performed by neutralization assay and titers are expressed in ED60.
  The analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies. The objective of this endpoint was to analyze the impact of the co-administration of RSVPreF3 with dTpa (Boostrix) (both formulations together) on the immunogenicity response to RSVPreF3.
Time Frame: At Day 8
Population: The analysis was performed on the PPS - Primary Study which consisted of all subjects from the ES - Primary Study, who complied with protocol defined procedures and for whom immunogenicity results were available for the specified assay and time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 98 | 99 | 100 | 102 | 100
Titers (ED60) | 14166 [12213 to 16431] | 14285 [11999 to 17008] | 10185 [8514 to 12183] | 10590 [8994 to 12469] | 783 [661 to 929]

11. Primary Outcome: RSV A Neutralizing Antibody GMTs at Day 31 [Primary Study]
Description: as for outcome 10
Time Frame: At Day 31
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 98 | 97 | 102 | 99 | 97
Titers (ED60) | 9836 [8252 to 11725] | 11038 [9160 to 13301] | 9214 [7806 to 10876] | 8739 [7561 to 10101] | 845 [705 to 1013]

12. Primary Outcome: RSV PreF3 IgG Antibody Geometric Mean Concentration (GMCs) at Screening [Primary Study]
Description: Serological assays for the determination of IgG antibodies against RSV PreF3 were performed by Enzyme-linked immunosorbent assay (ELISA ).
  The analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies. The objective of this endpoint was to analyze the impact of the co-administration of RSVPreF3 with dTpa (Boostrix) (both formulations together) on the immunogenicity response to RSVPreF3.
Time Frame: At Screening (Day -7 to Day 1)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units per milliliter (EU/mL)
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 100 | 100 | 103 | 102 | 102
ELISA Units per milliliter (EU/mL) | 6611 [5857 to 7461] | 6751 [5982 to 7620] | 7449 [6534 to 8492] | 6172 [5570 to 6840] | 6454 [5771 to 7217]

13. Primary Outcome: RSV PreF3 IgG GMCs at Day 8 [Primary Study]
Description: Serological assays for the determination of IgG antibodies against RSV PreF3 were performed by Enzyme-linked immunosorbent assay (ELISA).
  The analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies. The objective of this endpoint was to analyze the impact of the co-administration of RSVPreF3 with dTpa (Boostrix) (both formulations together) on the immunogenicity response to RSVPreF3.
Time Frame: At Day 8
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 99 | 99 | 100 | 102 | 100
EU/mL | 156568 [137244 to 178613] | 146708 [128639 to 167315] | 101662 [89783 to 115113] | 118670 [106004 to 132850] | 5780 [5145 to 6494]

14. Primary Outcome: RSV PreF3 IgG GMCs at Day 31 [Primary Study]
Description: Serological assays for the determination of IgG antibodies against RSV PreF3 were performed by Enzyme-linked immunosorbent assay (ELISA).
  Analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies. The objective of this endpoint was to analyze the impact of the co-administration of RSVPreF3 with dTpa (Boostrix) (both formulations together) on the immunogenicity response to RSVPreF3.
Time Frame: At Day 31
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 98 | 97 | 102 | 99 | 97
EU/mL | 101813 [89290 to 116092] | 106082 [93597 to 120231] | 86273 [77415 to 96145] | 88938 [79738 to 99200] | 6149 [5474 to 6908]

15. Secondary Outcome: Percentage of Subjects With Any Solicited Local Adverse Event (AEs) by Each Boostrix Formulation [Primary Study]
Description: Assessed solicited local AEs are: erythema, pain and swelling. Any = occurrence of the adverse event regardless of intensity grade. Any erythema and swelling = adverse event reported with a surface diameter greater than 0 millimeters.
  The analysis of this outcome measure was reported for each formulation of the dTpa (Boostrix) vaccine (300 μg or 500 μg of aluminum), as the objective of this endpoint was to analyze the impact of co-administration of RSVPreF3 with either 300 μg or 500 μg of dTpa (Boostrix) formulation on the safety response to RSVPreF3.
Time Frame: From Day 1 to Day 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- RSV120_dTpa_RSV120(EX-US): Subjects received one dose of 120 μg RSVPreF3 formulation 3 vaccine and one dose of 500 μg dTpa vaccine (Ex-US formulation) on Day 1 of the Primary Study and were followed up until Day 181. The subjects that agreed to participate in the Extension Study received a second dose of 120 μg RSVPreF3 formulation 3 vaccine (12 to 18 months post 1st vaccination) and were followed up until the study end.
- RSV120_Placebo_RSV120(EX-US); RSV120_Placebo_RSV120(US): Subjects received one dose of 120 μg RSVPreF3 formulation 3 vaccine and one dose of Placebo on Day 1 of the Primary Study and were followed up until Day 181. The subjects that agreed to participate in the Extension Study received a second dose of 120 μg RSVPreF3 formulation 3 vaccine 12 to 18 months post 1st vaccination and were followed up until the study end.
- RSV60_dTpa_RSV120(EX-US): Subjects received one dose of 60 μg RSVPreF3 formulation 2 vaccine and one dose of 500 μg dTpa vaccine (Ex-US formulation) on Day 1 of the Primary Study and were followed up until Day 181. The subjects that agreed to participate in the Extension Study received one dose of 120 μg RSVPreF3 formulation 3 vaccine 12 to 18 months post 1st vaccination and were followed up until the study end.
- RSV60_Placebo_RSV120(EX-US); RSV60_Placebo_RSV120(US): Subjects received one dose of 60 μg RSVPreF3 formulation 2 vaccine and one dose of Placebo on Day 1 of the Primary Study and were followed up until Day 181. The subjects that agreed to participate in the Extension Study received one dose of 120 μg RSVPreF3 formulation 3 vaccine 12 to 18 months post 1st vaccination and were followed up until the study end.
- dTpa_Placebo_RSV120(EX-US): Subjects received one dose of Placebo and one dose of 500 μg dTpa vaccine (Ex-US formulation) on Day 1 of the Primary Study and were followed up until Day 181. The subjects that agreed to participate in the Extension Study received one dose of 120 μg RSVPreF3 formulation 3 vaccine 12 to 18 months post 1st vaccination and were followed up until the study end.
- RSV120_dTpa_RSV120(US): Subjects received one dose of 120 μg RSVPreF3 formulation 3 vaccine and one dose of 300 μg dTpa vaccine (US formulation) on Day 1 of the Primary Study and were followed up until Day 181. The subjects that agreed to participate in the Extension Study received a second dose of 120 μg RSVPreF3 formulation 3 vaccine 12 to 18 months post 1st vaccination and were followed up until the study end.
- RSV60_dTpa_RSV120(US): Subjects received one dose of 60 μg RSVPreF3 formulation 2 vaccine and one dose of 300 μg dTpa vaccine (US formulation) on Day 1 of the Primary Study and were followed up until Day 181. The subjects that agreed to participate in the Extension Study received one dose of 120 μg RSVPreF3 formulation 3 vaccine 12 to 18 months post 1st vaccination and were followed up until the study end.
- dTpa_Placebo_RSV120(US): Subjects received one dose of Placebo and one dose of 300 μg dTpa vaccine (US formulation) on Day 1 of the Primary Study and were followed up until Day 181. The subjects that agreed to participate in the Extension Study received one dose of 120 μg RSVPreF3 formulation 3 vaccine 12 to 18 months post 1st vaccination and were followed up until the study end.
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV120_Placebo_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | RSV60_Placebo_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV120_Placebo_RSV120(US) | RSV60_dTpa_RSV120(US) | RSV60_Placebo_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 50 | 49 | 51 | 51 | 49 | 51 | 51 | 52 | 51 | 50
Percentage of participants
  Left Arm, Erythema | 6 [1.3 to 16.5] | 4.1 [0.5 to 14] | 5.9 [1.2 to 16.2] | 2 [0 to 10.4] | 0 [0 to 7.3] | 5.9 [1.2 to 16.2] | 5.9 [1.2 to 16.2] | 5.8 [1.2 to 15.9] | 9.8 [3.3 to 21.4] | 0 [0 to 7.1]
  Left Arm, Pain | 46 [31.8 to 60.7] | 53.1 [38.3 to 67.5] | 52.9 [38.5 to 67.1] | 60.8 [46.1 to 74.2] | 16.3 [7.3 to 29.7] | 56.9 [42.2 to 70.7] | 54.9 [40.3 to 68.9] | 51.9 [37.6 to 66] | 56.9 [42.2 to 70.7] | 22 [11.5 to 36]
  Left Arm, Swelling | 2 [0.1 to 10.6] | 6.1 [1.3 to 16.9] | 3.9 [0.5 to 13.5] | 2 [0 to 10.4] | 0 [0 to 7.3] | 2 [0 to 10.4] | 7.8 [2.2 to 18.9] | 1.9 [0 to 10.3] | 7.8 [2.2 to 18.9] | 0 [0 to 7.1]
  Right Arm, Erythema | 4 [0.5 to 13.7] | 2 [0.1 to 10.9] | 2 [0 to 10.4] | 2 [0 to 10.4] | 6.1 [1.3 to 16.9] | 3.9 [0.5 to 13.5] | 0 [0 to 7] | 7.7 [2.1 to 18.5] | 0 [0 to 7] | 6 [1.3 to 16.5]
  Right Arm, Pain | 86 [73.3 to 94.2] | 18.4 [8.8 to 32] | 88.2 [76.1 to 95.6] | 23.5 [12.8 to 37.5] | 79.6 [65.7 to 89.8] | 76.5 [62.5 to 87.2] | 31.4 [19.1 to 45.9] | 65.4 [50.9 to 78] | 13.7 [5.7 to 26.3] | 78 [64 to 88.5]
  Right Arm, Swelling | 6 [1.3 to 16.5] | 0 [0 to 7.3] | 3.9 [0.5 to 13.5] | 2 [0 to 10.4] | 6.1 [1.3 to 16.9] | 3.9 [0.5 to 13.5] | 0 [0 to 7] | 0 [0 to 6.8] | 0 [0 to 7] | 2 [0.1 to 10.6]

16. Secondary Outcome: Percentage of Subjects With Any Solicited General AEs by Each Boostrix Formulation [Primary Study]
Description: Assessed solicited general AEs are: fatigue, gastrointestinal symptoms, headache and fever(body temperature ≥ 38 degree celcius/100.4 degree Farenhit). Any = occurrence of the adverse event regardless of intensity grade or relation to study vaccination.
  The analysis of this outcome measure was reported for each formulation of the dTpa (Boostrix) vaccine (300 μg or 500 μg of aluminum), as the objective of this endpoint was to analyze the impact of co-administration of RSVPreF3 with either 300 μg or 500 μg of dTpa (Boostrix) formulation on the safety response to RSVPreF3.
Time Frame: From Day 1 to Day 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV120_Placebo_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | RSV60_Placebo_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV120_Placebo_RSV120(US) | RSV60_dTpa_RSV120(US) | RSV60_Placebo_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 50 | 49 | 51 | 51 | 49 | 51 | 52 | 52 | 51 | 50
Percentage of participants
  Fatigue | 36 [22.9 to 50.8] | 36.7 [23.4 to 51.7] | 39.2 [25.8 to 53.9] | 29.4 [17.5 to 43.8] | 34.7 [21.7 to 49.6] | 45.1 [31.1 to 59.7] | 42.3 [28.7 to 56.8] | 36.5 [23.6 to 51] | 35.3 [22.4 to 49.9] | 42 [28.2 to 56.8]
  Gastrointestinal symptoms | 22 [11.5 to 36] | 28.6 [16.6 to 43.3] | 23.5 [12.8 to 37.5] | 29.4 [17.5 to 43.8] | 30.6 [18.3 to 45.4] | 25.5 [14.3 to 39.6] | 28.8 [17.1 to 43.1] | 30.8 [18.7 to 45.1] | 27.5 [15.9 to 41.7] | 26 [14.6 to 40.3]
  Headache | 46 [31.8 to 60.7] | 38.8 [25.2 to 53.8] | 31.4 [19.1 to 45.9] | 45.1 [31.1 to 59.7] | 40.8 [27 to 55.8] | 43.1 [29.3 to 57.8] | 51.9 [37.6 to 66] | 38.5 [25.3 to 53] | 33.3 [20.8 to 47.9] | 34 [21.2 to 48.8]
  Temperature | 4 [0.5 to 13.7] | 6.1 [1.3 to 16.9] | 3.9 [0.5 to 13.5] | 5.9 [1.2 to 16.2] | 12.2 [4.6 to 24.8] | 0 [0 to 7] | 1.9 [0 to 10.3] | 1.9 [0 to 10.3] | 2 [0 to 10.4] | 2 [0.1 to 10.6]

17. Secondary Outcome: Percentage of Subjects With Any Unsolicited AEs by Each Boostrix Formulation [Primary Study]
Description: An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is to be reported as an unsolicited AE.
  The analysis of this outcome measure was reported for each formulation of the dTpa (Boostrix) vaccine (300 μg or 500 μg of aluminum), as the objective of this endpoint was to analyze the impact of co-administration of RSVPreF3 with either 300 μg or 500 μg of dTpa (Boostrix) formulation on the safety response to RSVPreF3.
Time Frame: From Day 1 to Day 31
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV120_Placebo_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | RSV60_Placebo_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV120_Placebo_RSV120(US) | RSV60_dTpa_RSV120(US) | RSV60_Placebo_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 50 | 49 | 51 | 51 | 51 | 51 | 52 | 52 | 51 | 51
Percentage of participants | 38 [24.7 to 52.8] | 36.7 [23.4 to 51.7] | 39.2 [25.8 to 53.9] | 43.1 [29.3 to 57.8] | 33.3 [20.8 to 47.9] | 39.2 [25.8 to 53.9] | 32.7 [20.3 to 47.1] | 26.9 [15.6 to 41] | 31.4 [19.1 to 45.9] | 31.4 [19.1 to 45.9]

18. Secondary Outcome: Number of Subjects With Any SAEs by Each Boostrix Formulation [Primary Study]
Description: A SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization or results in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study subject. Any is defined as any occurrence of SAE regardless of intensity grade or relation to study vaccination.
  The analysis of this outcome measure was reported for each formulation of the dTpa (Boostrix) vaccine (300 μg or 500 μg of aluminum), as the objective of this endpoint was to analyze the impact of co-administration of RSVPreF3 with either 300 μg or 500 μg of dTpa (Boostrix) formulation on the safety response to RSVPreF3.
Time Frame: From Day 1 to Day 31
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV120_Placebo_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | RSV60_Placebo_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV120_Placebo_RSV120(US) | RSV60_dTpa_RSV120(US) | RSV60_Placebo_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 50 | 49 | 51 | 51 | 51 | 51 | 52 | 52 | 51 | 51
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Subjects With Any SAEs From 1st Vaccination to Day 181 [Primary Study]
Description: as for outcome 4
Time Frame: From Day 1 to Day 181
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 101 | 101 | 103 | 102 | 102
Participants | 1 | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Subjects With Any SAEs From 1st Vaccination to Day 181 by Each Boostrix Formulation [Primary Study]
Description: as for outcome 18
Time Frame: From Day 1 to Day 181
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV120_Placebo_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | RSV60_Placebo_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV120_Placebo_RSV120(US) | RSV60_dTpa_RSV120(US) | RSV60_Placebo_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 50 | 49 | 51 | 51 | 51 | 51 | 52 | 52 | 51 | 51
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Subjects With Any SAEs From 2nd Vaccination to Day 181 Post 2nd Vaccination [Extension Period]
Description: A SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization or results in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study subject. Any is defined as any occurrence of SAE regardless of intensity grade or relation to study vaccination.
  The analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies, as the objective of this endpoint was to analyze the impact of the co-administration of RSVPreF3 with dTpa (Boostrix) (both formulations together) on the safety response to RSVPreF3.
Time Frame: From the Day of 2nd vaccination to Day 181 post 2nd vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 39 | 41 | 46 | 41 | 46
Participants | 0 | 0 | 0 | 1 | 0

22. Secondary Outcome: RSV A Neutralizing GMTs at Screening by Each Boostrix Formulation [Primary Study]
Description: Serological assays for the determination of antibodies against RSV-A were performed by neutralization assay and titers are expressed in ED60.
  The analysis of this outcome measure was reported for each formulation of the dTpa (Boostrix) vaccine (300 μg or 500 μg of aluminum), as the objective of this endpoint was to analyze the impact of co-administration of RSVPreF3 with either 300 μg or 500 μg of dTpa (Boostrix) formulation on the immunogenicity response to RSVPreF3.
Time Frame: At Screening (Day -7 to Day 1)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV120_Placebo_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | RSV60_Placebo_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV120_Placebo_RSV120(US) | RSV60_dTpa_RSV120(US) | RSV60_Placebo_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 49 | 49 | 51 | 51 | 51 | 51 | 51 | 52 | 51 | 51
Titers (ED60) | 777 [625 to 966] | 1009 [798 to 1277] | 989 [749 to 1307] | 777 [631 to 956] | 956 [740 to 1236] | 981 [773 to 1245] | 1035 [786 to 1362] | 1298 [1070 to 1574] | 765 [638 to 917] | 1154 [952 to 1399]

23. Secondary Outcome: RSV A Neutralizing GMTs at Day 8 by Each Boostrix Formulation [Primary Study]
Description: as for outcome 22
Time Frame: At Day 8
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV120_Placebo_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | RSV60_Placebo_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV120_Placebo_RSV120(US) | RSV60_dTpa_RSV120(US) | RSV60_Placebo_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 49 | 48 | 50 | 51 | 51 | 49 | 51 | 50 | 51 | 49
Titers (ED60) | 14523 [11831 to 17827] | 15458 [12424 to 19231] | 10677 [8146 to 13993] | 11128 [8885 to 13939] | 698 [530 to 918] | 13818 [11070 to 17248] | 13264 [10075 to 17462] | 9715 [7612 to 12400] | 10077 [7897 to 12858] | 884 [722 to 1082]

24. Secondary Outcome: RSV A Neutralizing GMTs at Day 31 by Each Boostrix Formulation [Primary Study]
Description: as for outcome 22
Time Frame: At Day 31
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV120_Placebo_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | RSV60_Placebo_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV120_Placebo_RSV120(US) | RSV60_dTpa_RSV120(US) | RSV60_Placebo_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 49 | 48 | 51 | 50 | 48 | 49 | 49 | 51 | 49 | 49
Titers (ED60) | 9838 [7987 to 12118] | 10800 [8675 to 13446] | 8754 [6821 to 11236] | 8141 [6545 to 10125] | 767 [575 to 1023] | 9834 [7354 to 13152] | 11276 [8283 to 15351] | 9698 [7735 to 12159] | 9395 [7726 to 11425] | 930 [740 to 1168]

25. Secondary Outcome: RSV A Neutralizing GMTs at Single Time Point Between 12 to 18 Months Post 1st Vaccination by Each Boostrix Formulation [Primary Study]
Description: as for outcome 22
Time Frame: At a single timepoint between 12 to 18 months post 1st vaccination
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV120_Placebo_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | RSV60_Placebo_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV120_Placebo_RSV120(US) | RSV60_dTpa_RSV120(US) | RSV60_Placebo_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 24 | 31 | 32 | 29 | 31 | 14 | 9 | 14 | 12 | 15
Titers (ED60) | 2034 [1458 to 2836] | 2869 [1998 to 4119] | 3086 [2143 to 4445] | 2200 [1522 to 3180] | 675 [495 to 920] | 2014 [1190 to 3411] | 2960 [1190 to 7362] | 2474 [1741 to 3517] | 2569 [1586 to 4160] | 969 [602 to 1560]

26. Secondary Outcome: RSV A Neutralizing GMTs at Single Time Point Between 12 to 18 Months Post 1st Vaccination [Primary Study]
Description: Serological assays for the determination of antibodies against RSV-A were performed by neutralization assay and titers are expressed in ED60.
  Analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies. The objective of this endpoint was to analyze the impact of the co-administration of RSVPreF3 with dTpa (Boostrix) (both formulations together) on the immunogenicity response to RSVPreF3.
Time Frame: At a single timepoint between 12 to 18 months post 1st vaccination
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 38 | 40 | 46 | 41 | 46
Titers (ED60) | 2027 [1546 to 2656] | 2889 [2086 to 4001] | 2885 [2204 to 3778] | 2302 [1730 to 3064] | 759 [588 to 980]

27. Secondary Outcome: RSV A Neutralizing GMTs at Day 31 Post 2nd Vaccination [Extension Study]
Description: Serological assays for the determination of antibodies against RSV-A were performed by neutralization assay and titers are expressed in ED60.
  The analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies, as the objective of this endpoint was to analyze the impact of the co-administration of RSVPreF3 with dTpa (Boostrix) (both formulations together) on the immunogenicity response to RSVPreF3.
Time Frame: At Day 31 post 2nd vaccination
Population: The analysis was performed on the PPS - Extension Study which consisted of all subjects from the ES - Extension Study, who complied with protocol defined procedures and for whom immunogenicity results were available for the specified assay and time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 38 | 37 | 44 | 39 | 42
Titers (ED60) | 3892 [3016 to 5022] | 5071 [3848 to 6683] | 4779 [3747 to 6094] | 4920 [3886 to 6231] | 8200 [6380 to 10539]

28. Secondary Outcome: RSV PreF3 IgG GMCs at Screening by Each Boostrix Formulation [Primary Study]
Description: Serological assays for the determination of IgG antibodies against RSV PreF3 were performed by ELISA. The corresponding antibody concentration is expressed in EU/mL. The cut-off value for the assay is 25 EU/mL.
  The analysis of this outcome measure was reported for each formulation of the dTpa (Boostrix) vaccine (300 μg or 500 μg of aluminum), as the objective of this endpoint was to analyze the impact of co-administration of RSVPreF3 with either 300 μg or 500 μg of dTpa (Boostrix) formulation on the immunogenicity response to RSVPreF3.
Time Frame: At Screening (Day -7 to Day 1)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV120_Placebo_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | RSV60_Placebo_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV120_Placebo_RSV120(US) | RSV60_dTpa_RSV120(US) | RSV60_Placebo_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 49 | 49 | 51 | 51 | 51 | 51 | 51 | 52 | 51 | 51
EU/mL | 6240 [5159 to 7548] | 6524 [5597 to 7604] | 7237 [5905 to 8869] | 6106 [5275 to 7067] | 5907 [5077 to 6873] | 6987 [5975 to 8170] | 6978 [5764 to 8447] | 7662 [6447 to 9107] | 6240 [5375 to 7245] | 7051 [5973 to 8324]

29. Secondary Outcome: RSV PreF3 IgG GMCs at Day 8 by Each Boostrix Formulation [Primary Study]
Description: Serological assays for the determination of IgG antibodies against RSV PreF3 were performed by ELISA. The corresponding antibody concentration is expressed in EU/mL. The cut-off value for the assay is 25 EU/mL. The analysis of this outcome measure was reported for each formulation of the Boostrix (300 μg or 500 μg of aluminum). The objective of this endpoint was to analyze the impact of co-administration of RSVPreF3 with either 300 μg or 500 μg of Boostrix formulation on the immunogenicity response to RSVPreF3.
Time Frame: At Day 8
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV120_Placebo_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | RSV60_Placebo_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV120_Placebo_RSV120(US) | RSV60_dTpa_RSV120(US) | RSV60_Placebo_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 49 | 48 | 50 | 51 | 51 | 50 | 51 | 50 | 51 | 49
EU/mL | 155721 [133435 to 181728] | 143104 [126138 to 162352] | 100064 [84699 to 118216] | 123475 [107405 to 141950] | 5523 [4700 to 6490] | 157403 [126554 to 195772] | 150184 [119250 to 189142] | 103286 [85400 to 124919] | 114053 [95089 to 136799] | 6061 [5097 to 7207]

30. Secondary Outcome: RSV PreF3 IgG GMCs at Day 31 by Each Boostrix Formulation [Primary Study]
Description: as for outcome 28
Time Frame: At Day 31
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV120_Placebo_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | RSV60_Placebo_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV120_Placebo_RSV120(US) | RSV60_dTpa_RSV120(US) | RSV60_Placebo_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 49 | 48 | 51 | 50 | 48 | 49 | 49 | 51 | 49 | 49
EU/mL | 94254 [80742 to 110026] | 95113 [83282 to 108624] | 84509 [72281 to 98805] | 81915 [70291 to 95460] | 5600 [4777 to 6565] | 109978 [88643 to 136446] | 118052 [95525 to 145892] | 88075 [75406 to 102872] | 96727 [82608 to 113258] | 6739 [5678 to 7999]

31. Secondary Outcome: RSV PreF3 IgG GMCs at Single Time Point Between 12 to 18 Months Post 1st Vaccination by Each Boostrix Formulation [Primary Study]
Description: as for outcome 29
Time Frame: At a single timepoint between 12 to 18 months post 1st vaccination
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV120_Placebo_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | RSV60_Placebo_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV120_Placebo_RSV120(US) | RSV60_dTpa_RSV120(US) | RSV60_Placebo_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 24 | 31 | 32 | 29 | 31 | 14 | 9 | 14 | 12 | 15
EU/mL | 18832 [15141 to 23423] | 20894 [16466 to 26512] | 23189 [18629 to 28864] | 20720 [16689 to 25726] | 5014 [3932 to 6392] | 18127 [10969 to 29958] | 19641 [9143 to 42195] | 22905 [17801 to 29471] | 22233 [15931 to 31029] | 6811 [5005 to 9269]

32. Secondary Outcome: RSV PreF3 IgG GMCs at Single Time Point Between 12 to 18 Months Post 1st Vaccination [Primary Study]
Description: Serological assays for the determination of IgG antibodies against RSV PreF3 were performed by ELISA. The corresponding antibody concentration is expressed in EU/mL. The cut-off value for the assay is 25 EU/mL.
  Analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies. The objective of this endpoint was to analyze the impact of the co-administration of RSVPreF3 with dTpa (Boostrix) (both formulations together) on the immunogenicity response to RSVPreF3.
Time Frame: At a single timepoint between 12 to 18 months post 1st vaccination
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 38 | 40 | 46 | 41 | 46
EU/mL | 18570 [14961 to 23049] | 20605 [16333 to 25995] | 23102 [19586 to 27249] | 21152 [17777 to 25168] | 5540 [4581 to 6700]

33. Secondary Outcome: RSV PreF3 IgG GMCs at Day 31 Post 2nd Vaccination [Extension Study]
Description: Serological assays for the determination of IgG antibodies against RSV PreF3 were performed by ELISA.
  The analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies, as the objective of this endpoint was to analyze the impact of the co-administration of RSVPreF3 with dTpa (Boostrix) (both formulations together) on the immunogenicity response to RSVPreF3.
Time Frame: At Day 31 post 2nd vaccination
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: (IU/mL)
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 38 | 37 | 44 | 39 | 42
(IU/mL) | 41399 [34806 to 49241] | 42943 [37226 to 49537] | 43977 [38784 to 49865] | 45680 [38574 to 54094] | 86934 [75442 to 100177]

34. Secondary Outcome: Pertussis Toxoid (Anti-PT), Filamentous Hemagglutinin (Anti-FHA) and Pertactin (Anti-PRN) GMCs at Screening by Each Boostrix Formulation [Primary Study]
Description: Serological assays for the determination of IgG antibodies against Bordetella pertussis: anti-PT, anti-FHA and anti-PRN were performed by ELISA.
  The analysis of this outcome measure was reported for each formulation of the dTpa (Boostrix) vaccine (300 μg or 500 μg of aluminum).
Time Frame: At Screening (Day -7 to Day 1)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: International Units Per mL (IU/mL)
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV60_dTpa_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 49 | 51 | 51 | 51 | 52 | 51
International Units Per mL (IU/mL)
  anti-PT | 7.39 [5.11 to 10.68] | 7.64 [5.47 to 10.66] | 6.65 [4.66 to 9.47] | 7.55 [5.34 to 10.66] | 5.66 [4.06 to 7.88] | 7.17 [4.94 to 10.41]
  anti-FHA | 32.8 [23 to 46.7] | 34.5 [24.3 to 49.1] | 29.3 [22 to 38.9] | 31 [22.7 to 42.4] | 29.6 [22.5 to 38.9] | 28 [21 to 37.4]
  anti-PRN | 43.2 [27.9 to 66.7] | 39 [25.3 to 60.1] | 28.1 [18.2 to 43.4] | 42.1 [27.6 to 64.2] | 40.1 [26.9 to 60] | 28.7 [17.9 to 46.1]

35. Secondary Outcome: Pertussis Toxoid (Anti-PT), Filamentous Hemagglutinin (Anti-FHA) and Pertactin (Anti-PRN) GMCs at Day 31 by Each Boostrix Formulation [Primary Study]
Description: as for outcome 34
Time Frame: At Day 31
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: (IU/mL)
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV60_dTpa_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 49 | 51 | 48 | 49 | 51 | 49
(IU/mL)
  anti-PT | 57.36 [41.82 to 78.69] | 54.95 [44.78 to 67.44] | 79.16 [62.67 to 99.98] | 43.76 [34.1 to 56.17] | 36.98 [28.25 to 48.42] | 44.99 [34.81 to 58.15]
  anti-FHA | 237.1 [194.1 to 289.5] | 210.6 [168.5 to 263.1] | 303.6 [241.6 to 381.5] | 186.5 [149.8 to 232.3] | 176.7 [139.3 to 224.1] | 232.9 [182.2 to 297.8]
  anti-PRN: number analyzed (Participants) | 49 | 51 | 47 | 49 | 51 | 49
  anti-PRN | 309.5 [226.7 to 422.6] | 214.7 [166.8 to 276.4] | 395.1 [290.3 to 537.6] | 217.7 [153.7 to 308.3] | 228.1 [161.9 to 321.5] | 331.4 [238.4 to 460.5]

36. Secondary Outcome: Diphtheria (Anti-D) GMC at Screening by Each Boostrix Formulation [Primary Study]
Description: Serological assays for the determination of IgG antibodies against anti-D were performed by ELISA.
  The analysis of this outcome measure was reported for each formulation of the dTpa (Boostrix) vaccine (300 μg or 500 μg of aluminum).
Time Frame: At Screening (Day -7 to Day 1)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: (IU/mL)
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV60_dTpa_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 49 | 51 | 49 | 49 | 52 | 50
(IU/mL) | 0.26 [0.18 to 0.39] | 0.27 [0.17 to 0.42] | 0.23 [0.16 to 0.32] | 0.46 [0.33 to 0.64] | 0.55 [0.42 to 0.73] | 0.58 [0.43 to 0.78]

37. Secondary Outcome: Diphtheria (Anti-D) GMCs at Day 31 by Each Boostrix Formulation [Primary Study]
Description: as for outcome 36
Time Frame: At Day 31
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: (IU/mL)
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV60_dTpa_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 49 | 51 | 48 | 47 | 48 | 49
(IU/mL) | 1.3 [0.97 to 1.73] | 1.18 [0.85 to 1.63] | 1.76 [1.25 to 2.48] | 2.11 [1.61 to 2.76] | 2.2 [1.72 to 2.81] | 3.29 [2.62 to 4.14]

38. Secondary Outcome: Tetanus (Anti-T) GMCs at Screening by Each Boostrix Formulation [Primary Study]
Description: Serological assays for the determination of IgG antibodies against anti-T were performed by ELISA.
  The analysis of this outcome measure was reported for each formulation of the dTpa (Boostrix) vaccine (300 μg or 500 μg of aluminum).
Time Frame: At Screening (Day -7 to Day 1)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: (IU/mL)
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV60_dTpa_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 49 | 51 | 51 | 51 | 52 | 51
(IU/mL) | 1.14 [0.87 to 1.5] | 1.1 [0.78 to 1.54] | 0.88 [0.64 to 1.22] | 1.35 [1.01 to 1.81] | 1.56 [1.27 to 1.92] | 1.68 [1.29 to 2.19]

39. Secondary Outcome: Tetanus (Anti-T) GMCs at Day 31 by Each Boostrix Formulation [Primary Study]
Description: as for outcome 38
Time Frame: At Day 31
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: (IU/mL)
Arm/Group | RSV120_dTpa_RSV120(EX-US) | RSV60_dTpa_RSV120(EX-US) | dTpa_Placebo_RSV120(EX-US) | RSV120_dTpa_RSV120(US) | RSV60_dTpa_RSV120(US) | dTpa_Placebo_RSV120(US)
Number analyzed (Participants) | 49 | 51 | 48 | 49 | 51 | 49
(IU/mL) | 5.57 [4.64 to 6.7] | 5.3 [4.52 to 6.21] | 6.74 [5.79 to 7.84] | 6.09 [4.98 to 7.45] | 6.27 [5.29 to 7.44] | 8.32 [6.88 to 10.05]

40. Secondary Outcome: Pertussis Toxoid (Anti-PT), Filamentous Hemagglutinin (Anti-FHA) and Pertactin (Anti-PRN) GMCs at Screening [Primary Study]
Description: Serological assays for the determination of IgG antibodies against Bordetella pertussis: anti-PT, anti-FHA and anti-PRN were performed by ELISA.
  Analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies.
Time Frame: At Screening (Day -7 to Day 1)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 100 | 103 | 102
IU/mL
  Anti-PT | 7.47 [5.83 to 9.57] | 6.56 [5.20 to 8.28] | 6.90 [5.36 to 8.89]
  Anti-FHA | 31.9 [25.3 to 40.2] | 31.9 [25.6 to 39.8] | 28.6 [23.5 to 34.9]
  Anti-PRN | 42.6 [31.6 to 57.4] | 39.6 [29.6 to 52.9] | 28.4 [20.7 to 38.9]

41. Secondary Outcome: Pertussis Toxoid (Anti-PT), Filamentous Hemagglutinin (Anti-FHA) and Pertactin (Anti-PRN) GMCs at Day 31 [Primary Study]
Description: as for outcome 40
Time Frame: At Day 31
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 98 | 102 | 97
IU/mL
  Anti-PT | 50.10 [41.04 to 61.17] | 45.08 [38.00 to 53.48] | 59.51 [49.71 to 71.23]
  Anti-FHA | 210.3 [181.4 to 243.8] | 192.9 [164.2 to 226.6] | 265.6 [224.7 to 313.8]
  Anti-PRN: number analyzed (Participants) | 98 | 102 | 96
  Anti-PRN | 259.6 [205.8 to 327.4] | 221.3 [179.5 to 272.9] | 361.1 [289.1 to 451.1]

42. Secondary Outcome: Diphtheria (Anti-D) GMCs at Screening [Primary Study]
Description: Serological assays for the determination of IgG antibodies against anti-D were performed by ELISA.
  Analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies.
Time Frame: At Screening (Day -7 to Day 1)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 98 | 103 | 99
IU/mL | 0.35 [0.27 to 0.45] | 0.39 [0.30 to 0.51] | 0.36 [0.28 to 0.47]

43. Secondary Outcome: Diphtheria (Anti-D) GMCs at Day 31 [Primary Study]
Description: as for outcome 42
Time Frame: At Day 31
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 96 | 99 | 97
IU/mL | 1.65 [1.35 to 2.01] | 1.59 [1.29 to 1.97] | 2.42 [1.96 to 2.99]

44. Secondary Outcome: Tetanus (Anti-T) GMCs at Screening [Primary Study]
Description: Serological assays for the determination of IgG antibodies against anti-T were performed by ELISA.
  Analysis of this outcome measure was reported for the Pooled groups [RSV120_dTpa_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled) and dTpa_Placebo_RSV120(Pooled)] as the two formulations of the dTpa vaccine (containing 300 μg or 500 μg of aluminum) showed similar immunogenicity and safety profiles in previous studies.
Time Frame: At Screening (Day -7 to Day 1)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 100 | 103 | 102
IU/mL | 1.24 [1.02 to 1.51] | 1.31 [1.08 to 1.60] | 1.22 [0.98 to 1.51]

45. Secondary Outcome: Tetanus (Anti-T) GMCs at Day 31 [Primary Study]
Description: as for outcome 44
Time Frame: At Day 31
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
Number analyzed (Participants) | 98 | 102 | 97
IU/mL | 5.83 [5.10 to 6.66] | 5.76 [5.13 to 6.47] | 7.49 [6.64 to 8.46]

ADVERSE EVENTS:
Time Frame: Solicited adverse events were collected during the 7-day follow-up period and unsolicited adverse events during the 30-day follow-up period after any vaccination. Serious adverse events were collected from Day 1 (Primary Study) to the Study End (Day 181 after the second RSVPreF3 vaccination, Extension Study).
Description: As per the analysis plan, AEs were reported for the RSV120_dTpa_RSV120(Pooled), RSV120_Placebo_RSV120(Pooled), RSV60_dTpa_RSV120(Pooled), RSV60_Placebo_RSV120(Pooled) & dTpa_Placebo_RSV120(Pooled) groups, as the 2 formulations of dTpa vaccine (300 μg/500 μg) showed similar safety profiles in previous studies.Total number of subjects affected by Other AEs were obtained from the rows with the maximum number of events.Results of Other AEs were summarized by two periods (Primary & Extension Study).
Arm/Group | RSV120_dTpa_RSV120(Pooled) | RSV120_Placebo_RSV120(Pooled) | RSV60_dTpa_RSV120(Pooled) | RSV60_Placebo_RSV120(Pooled) | dTpa_Placebo_RSV120(Pooled)
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/101 | 0/103 | 0/102 | 0/102
Serious Adverse Events (participants affected / at risk) | 1/101 | 0/101 | 0/103 | 1/102 | 0/102
Other Adverse Events (participants affected / at risk) | 92/101 | 90/101 | 91/103 | 82/102 | 89/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV120_dTpa_RSV120(Pooled) (N=101) | RSV120_Placebo_RSV120(Pooled) (N=101) | RSV60_dTpa_RSV120(Pooled) (N=103) | RSV60_Placebo_RSV120(Pooled) (N=102) | dTpa_Placebo_RSV120(Pooled) (N=102)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | RSV120_dTpa_RSV120(Pooled) (N=101) | RSV120_Placebo_RSV120(Pooled) (N=101) | RSV60_dTpa_RSV120(Pooled) (N=103) | RSV60_Placebo_RSV120(Pooled) (N=102) | dTpa_Placebo_RSV120(Pooled) (N=102)
Injection site pain - Primary Study (General disorders) | 86 (204) | 62 (136) | 84 (200) | 60 (128) | 81 (170)
Fatigue - Primary Study (General disorders) | 42 (86) | 40 (83) | 39 (79) | 34 (69) | 38 (77)
Injection site erythema - Primary Study (General disorders) | 7 (18) | 6 (12) | 8 (18) | 7 (14) | 6 (12)
Injection site swelling - Primary Study (General disorders) | 5 (12) | 8 (16) | 3 (6) | 6 (12) | 4 (8)
Pyrexia - Primary Study (General disorders) | 2 (4) | 4 (8) | 3 (6) | 4 (8) | 7 (14)
Injection site bruising - Primary Study (General disorders) | 2 (4) | 2 (6) | 4 (8) | 1 (2) | 2 (4)
Administration site pain - Primary Study (General disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Administration site erythema - Primary Study (General disorders) | 0 (0) | 3 (3) | 4 (4) | 1 (1) | 0 (0)
Injection site pruritus - Primary Study (General disorders) | 1 (2) | 2 (4) | 0 (0) | 1 (2) | 3 (6)
Administration site swelling - Primary Study (General disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Injection site haemorrhage - Primary Study (General disorders) | 0 (0) | 2 (4) | 1 (2) | 1 (2) | 0 (0)
Vaccination site nodule - Primary Study (General disorders) | 1 (2) | 0 (0) | 2 (4) | 0 (0) | 1 (2)
Malaise - Primary Study (General disorders) | 1 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Pain - Primary Study (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Injection site warmth - Primary Study (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (4)
Axillary pain - Primary Study (General disorders) | 1 (2) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Chills - Primary Study (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Injection site induration - Primary Study (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Influenza like illness - Primary Study (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Feeling cold - Primary Study (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hangover - Primary Study (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site discomfort - Primary Study (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma - Primary Study (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site discolouration - Primary Study (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Injection site rash - Primary Study (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Headache - Primary Study (Nervous system disorders) | 47 (105) | 47 (101) | 38 (81) | 42 (92) | 37 (76)
Dizziness - Primary Study (Nervous system disorders) | 2 (4) | 2 (4) | 0 (0) | 1 (2) | 1 (2)
Disturbance in attention - Primary Study (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine - Primary Study (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sciatica - Primary Study (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort - Primary Study (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neuralgia - Primary Study (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sleep deficit - Primary Study (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Post-traumatic headache - Primary Study (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal disorder - Primary Study (Gastrointestinal disorders) | 24 (50) | 29 (60) | 28 (57) | 29 (58) | 28 (56)
Nausea - Primary Study (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Dyspepsia - Primary Study (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Toothache - Primary Study (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Abdominal distension - Primary Study (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea - Primary Study (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperchlorhydria - Primary Study (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain - Primary Study (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection - Primary Study (Infections and infestations) | 8 (16) | 9 (18) | 4 (8) | 2 (4) | 5 (10)
Nasopharyngitis - Primary Study (Infections and infestations) | 1 (2) | 1 (2) | 0 (0) | 7 (14) | 3 (6)
Urinary tract infection - Primary Study (Infections and infestations) | 1 (2) | 0 (0) | 1 (2) | 1 (2) | 2 (4)
Sinusitis - Primary Study (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 2 (4)
Rhinitis - Primary Study (Infections and infestations) | 1 (2) | 1 (2) | 0 (0) | 1 (2) | 1 (2)
Gastroenteritis - Primary Study (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 2 (4) | 1 (2)
Pharyngitis - Primary Study (Infections and infestations) | 1 (2) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Tooth infection - Primary Study (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Conjunctivitis - Primary Study (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis bacterial - Primary Study (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal - Primary Study (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Viral infection - Primary Study (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis - Primary Study (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Chlamydial infection - Primary Study (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cystitis - Primary Study (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ear infection - Primary Study (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gingivitis - Primary Study (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oral herpes - Primary Study (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Otitis media - Primary Study (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Otitis media acute - Primary Study (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vaginitis chlamydial - Primary Study (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection - Primary Study (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myalgia - Primary Study (Musculoskeletal and connective tissue disorders) | 2 (4) | 4 (8) | 1 (2) | 4 (8) | 0 (0)
Back pain - Primary Study (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 1 (2) | 2 (4) | 2 (4)
Neck pain - Primary Study (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Arthralgia - Primary Study (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (4) | 0 (0)
Muscle tightness - Primary Study (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity - Primary Study (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Musculoskeletal pain - Primary Study (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness - Primary Study (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pain in jaw - Primary Study (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Oropharyngeal pain - Primary Study (Respiratory, thoracic and mediastinal disorders) | 3 (8) | 2 (4) | 1 (2) | 1 (2) | 0 (0)
Cough - Primary Study (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (2) | 2 (4) | 0 (0)
Rhinorrhoea - Primary Study (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Nasal congestion - Primary Study (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Rash - Primary Study (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (2)
Dermatitis - Primary Study (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic - Primary Study (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats - Primary Study (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lymphadenopathy - Primary Study (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 2 (4) | 2 (4) | 0 (0)
Lymphadenitis - Primary Study (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain - Primary Study (Injury, poisoning and procedural complications) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Thermal burn - Primary Study (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dysmenorrhoea - Primary Study (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Intermenstrual bleeding - Primary Study (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vaginal discharge - Primary Study (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Insomnia - Primary Study (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (2) | 0 (0)
Drug hypersensitivity - Primary Study (Immune system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations - Primary Study (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Injection site pain - Extension Study (General disorders) | 34/39 (68) | 36/41 (74) | 37/46 (74) | 35/41 (70) | 18/46 (38)
Fatigue - Extension Study (General disorders) | 10/39 (23) | 15/41 (31) | 17/46 (35) | 19/41 (39) | 16/46 (32)
Injection site erythema - Extension Study (General disorders) | 7/39 (14) | 4/41 (8) | 4/46 (8) | 6/41 (12) | 1/46 (2)
Injection site swelling - Extension Study (General disorders) | 5/39 (10) | 3/41 (6) | 4/46 (8) | 2/41 (4) | 1/46 (2)
Pyrexia - Extension Study (General disorders) | 0/39 (0) | 0/41 (0) | 1/46 (2) | 5/41 (10) | 1/46 (2)
Injection site pruritus - Extension Study (General disorders) | 0/39 (0) | 1/41 (2) | 0/46 (0) | 2/41 (4) | 0/46 (0)
Malaise - Extension Study (General disorders) | 1/39 (2) | 0/41 (0) | 1/46 (2) | 0/41 (0) | 0/46 (0)
Administration site pain - Extension Study (General disorders) | 1/39 (1) | 0/41 (0) | 0/46 (0) | 0/41 (0) | 0/46 (0)
Injection site induration - Extension Study (General disorders) | 1/39 (2) | 0/41 (0) | 0/46 (0) | 0/41 (0) | 0/46 (0)
Inflammation - Extension Study (General disorders) | 0/39 (0) | 1/41 (2) | 0/46 (0) | 0/41 (0) | 0/46 (0)
Influenza like illness - Extension Study (General disorders) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 1/41 (2) | 0/46 (0)
Injection site haemorrhage - Extension Study (General disorders) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 1/41 (2) | 0/46 (0)
Pain - Extension Study (General disorders) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 1/41 (2) | 0/46 (0)
Administration site swelling - Extension Study (General disorders) | 0/39 (0) | 0/41 (0) | 1/46 (1) | 0/41 (0) | 0/46 (0)
Injection site lymphadenopathy - Extension Study (General disorders) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 0/41 (0) | 1/46 (2)
Headache - Extension Study (Nervous system disorders) | 11/39 (24) | 15/41 (31) | 15/46 (32) | 23/41 (50) | 16/46 (34)
Migraine with aura - Extension Study (Nervous system disorders) | 0/39 (0) | 0/41 (0) | 1/46 (2) | 0/41 (0) | 0/46 (0)
Gastrointestinal disorder - Extension Study (Gastrointestinal disorders) | 4/39 (9) | 10/41 (20) | 7/46 (14) | 10/41 (20) | 7/46 (14)
Oesophageal spasm - Extension Study (Gastrointestinal disorders) | 0/39 (0) | 0/41 (0) | 1/46 (2) | 0/41 (0) | 1/46 (2)
Abdominal pain - Extension Study (Gastrointestinal disorders) | 1/39 (2) | 0/41 (0) | 0/46 (0) | 0/41 (0) | 0/46 (0)
Diarrhoea - Extension Study (Gastrointestinal disorders) | 1/39 (2) | 0/41 (0) | 0/46 (0) | 0/41 (0) | 0/46 (0)
Vomiting - Extension Study (Gastrointestinal disorders) | 1/39 (2) | 0/41 (0) | 0/46 (0) | 0/41 (0) | 0/46 (0)
Pharyngitis - Extension Study (Infections and infestations) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 2/41 (4) | 0/46 (0)
Nasopharyngitis - Extension Study (Infections and infestations) | 0/39 (0) | 0/41 (0) | 1/46 (2) | 1/41 (2) | 0/46 (0)
Bronchitis - Extension Study (Infections and infestations) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 1/41 (2) | 0/46 (0)
Ear infection - Extension Study (Infections and infestations) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 1/41 (2) | 0/46 (0)
Gastroenteritis - Extension Study (Infections and infestations) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 1/41 (2) | 0/46 (0)
Pyelonephritis - Extension Study (Infections and infestations) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 1/41 (1) | 0/46 (0)
Tonsillitis - Extension Study (Infections and infestations) | 0/39 (0) | 1/41 (2) | 0/46 (0) | 0/41 (0) | 0/46 (0)
Respiratory tract infection - Extension Study (Infections and infestations) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 0/41 (0) | 1/46 (2)
Sinusitis - Extension Study (Infections and infestations) | 0/39 (0) | 0/41 (0) | 1/46 (2) | 0/41 (0) | 0/46 (0)
Upper respiratory tract infection - Extension Study (Infections and infestations) | 0/39 (0) | 0/41 (0) | 1/46 (2) | 0/41 (0) | 0/46 (0)
Oropharyngeal pain - Extension Study (Respiratory, thoracic and mediastinal disorders) | 0/39 (0) | 3/41 (6) | 1/46 (2) | 0/41 (0) | 0/46 (0)
Nasal congestion - Extension Study (Respiratory, thoracic and mediastinal disorders) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 1/41 (2) | 0/46 (0)
Rhinorrhoea - Extension Study (Respiratory, thoracic and mediastinal disorders) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 0/41 (0) | 1/46 (2)
Limb discomfort - Extension Study (Musculoskeletal and connective tissue disorders) | 1/39 (2) | 0/41 (0) | 0/46 (0) | 0/41 (0) | 1/46 (2)
Myalgia - Extension Study (Musculoskeletal and connective tissue disorders) | 0/39 (0) | 1/41 (2) | 0/46 (0) | 0/41 (0) | 1/46 (2)
Arthralgia - Extension Study (Musculoskeletal and connective tissue disorders) | 1/39 (2) | 0/41 (0) | 0/46 (0) | 0/41 (0) | 0/46 (0)
Muscle strain - Extension Study (Injury, poisoning and procedural complications) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 1/41 (2) | 0/46 (0)
Contusion - Extension Study (Injury, poisoning and procedural complications) | 0/39 (0) | 0/41 (0) | 1/46 (2) | 0/41 (0) | 0/46 (0)
Affect lability - Extension Study (Psychiatric disorders) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 1/41 (2) | 0/46 (0)
Poor quality sleep - Extension Study (Psychiatric disorders) | 0/39 (0) | 0/41 (0) | 1/46 (2) | 0/41 (0) | 0/46 (0)
Night sweats - Extension Study (Skin and subcutaneous tissue disorders) | 0/39 (0) | 1/41 (2) | 0/46 (0) | 0/41 (0) | 0/46 (0)
Rash - Extension Study (Skin and subcutaneous tissue disorders) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 0/41 (0) | 1/46 (2)
Ear pain - Extension Study (Ear and labyrinth disorders) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 1/41 (2) | 0/46 (0)
Dysmenorrhoea - Extension Study (Reproductive system and breast disorders) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 1/41 (2) | 0/46 (0)
Vision blurred - Extension Study (Eye disorders) | 0/39 (0) | 0/41 (0) | 1/46 (2) | 0/41 (0) | 0/46 (0)
Seasonal allergy - Extension Study (Immune system disorders) | 0/39 (0) | 0/41 (0) | 1/46 (2) | 0/41 (0) | 0/46 (0)
Hypertension - Extension Study (Vascular disorders) | 0/39 (0) | 0/41 (0) | 0/46 (0) | 0/41 (0) | 1/46 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT04138056/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/56/NCT04138056/SAP_001.pdf